CLINICAL TRIAL: NCT03604796
Title: Alternative Acetaminophen Treatment of the Hemodynamivally Significant Patent Ductus Arteriosus in Preterm Neonates Who Are Not Candidates for Enteral Administration: A Pilot Study
Brief Title: Alternative Paracetamol Treatments for the Neonate With a hsPDA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0207-18-SZMC
Record Dates: First submitted 2018-07-19; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Ductus Arteriosus, Patent
Keywords: acetaminophen
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Acetaminophen; Infusions, Intravenous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous IV Acetaminophen (Active Comparator): Intravenous Infusion
  Interventions: Drug: Intravenous Infusion
- Rectal Acetaminophen (Active Comparator): Rectal Solution
  Interventions: Drug: Rectal Solution

INTERVENTIONS:
Drug: Rectal Solution — Rectal acetaminophen at 15 mg/kg x 4/day for three days
  Other Names: acetaminophen / paracetamol
  Arms: Rectal Acetaminophen
Drug: Intravenous Infusion — Loading dose of 15 mg/kg IV acetaminophen followed by a continuous infusion at a rate of 2.5 mg/kg/hr for 72 hours
  Other Names: acetaminophen / paracetamol
  Arms: Continuous IV Acetaminophen

SUMMARY:
Early targeted treatment of a hemodynamically significant patent ductus arteriosus (hsPDA) during the first week of life in preterm neonates is often recommended. Our standard first line therapeutic approach is enteral acetaminophen. However many extremely low birth weight infants may be on limited or no feeds when PDA closure is determined to be indicated, thus restricting the use of enteral acetaminophen. Several studies have suggested that intravenous acetaminophen is less effective than enteral. Thus, in this study, we propose to compare two alternative modes of administration when enteral acetaminophen is not an option.

DETAILED DESCRIPTION:
Once parental consent for entrance into the study is obtained, eligible babies will be randomized to receive either IV acetaminophen (perfalgen) by continuous infusion at 2.5 mg/kg/h following a loading dose of 15 mg /kg/ over 20 minutes or rectal acetaminophen at 15 mg/kg every 6 hours for a period of 3 days.

ELIGIBILITY:
Inclusion Criteria:

Inborn preterm neonates, < 1000 gm birth weight; < 28 weeks' gestational age; who are admitted to the neonatal intensive care unit of the Shaare Zedek Medical Center and are diagnosed with a hemodynamically significant patent ductus arteriosus within the first week of life and who are on limited or no enteral feeds -

Exclusion Criteria:

Other congenital heart disease, major congenital anomalies, sepsis; and/or NEC.

Ages: 2 Days to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Ductal closure | Up to 1 week following treatment
  Follow-up echocardiogram showing closed ductus arteriosus

SECONDARY OUTCOMES:
PDA Ligation | Completion of study intervention until 40 weeks post-conception
  Need for surgical ligation

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Hammerman, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Neonatal Intensive Care Unit - Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No